CLINICAL TRIAL: NCT02295540
Title: Preoperative Hypofractionated Radiation Followed by Surgery in Advanced Oral Cavity Squamous Cell Carcinoma
Brief Title: Hypofractionated Radiation Therapy Followed by Surgery in Treating Patients With Advanced Squamous Cell Carcinoma of the Oral Cavity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Sung Kim, MD, Residency and Clinical Director, Residency Director, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro20140000684; NCI-2014-02215 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 031401 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Tongue Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Preoperative hypofractionated radiation followed by surgical resection
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (hypofractionated IMRT, surgery) (Experimental): Patients undergo hypofractionated IMRT every other day for up to 5 treatments. Patients then undergo surgery 7-14 days after the last radiation treatment.
  Interventions: Radiation: hypofractionated radiation therapy; Radiation: intensity-modulated radiation therapy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: hypofractionated radiation therapy — Undergo hypofractionated IMRT
Radiation: intensity-modulated radiation therapy — Undergo hypofractionated IMRT
  Other Names: IMRT
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies how well hypofractionated radiation therapy followed by surgery works in treating patients with squamous cell carcinoma of the oral cavity that has spread to other places in the body. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Giving hypofractionated radiation therapy before surgery may shrink the tumor making it easier to be removed, may reduce the risk of the cancer coming back, and may be a better treatment for squamous cell carcinoma of the oral cavity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. 2 year locoregional control for advanced oral cavity squamous cell carcinoma (SCC) treated with preoperative hypofractionated radiation followed by surgical resection.

SECONDARY OBJECTIVES:

I. Rate of pathologic complete response after preoperative hypofractionated radiation at both the primary site and lymph nodes (LN).

II. Rate of radiologic complete and partial response (computed tomography [CT] neck with intravenous [IV] contrast performed before and after radiation therapy, judged per Response Evaluation Criteria In Solid Tumors [RECIST] 1.1 criteria).

III. Grade III/IV/V toxicity both short term (from start of radiation to 60 days after surgery) and long term (more than 60 days after surgery).

IV. Rate of flap complications: Rate of flap revisions, and complete revisions required.

V. Molecular correlates. VI. Quantitative imaging correlates.

OUTLINE:

Patients undergo hypofractionated intensity-modulated radiation therapy (IMRT) every other day for up to 5 treatments. Patients then undergo surgery 7-14 days after the last radiation treatment.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to sign study specific informed consent
* Pathologically proven (histologically or cytologically) diagnosis of squamous cell carcinoma (including histological variants like papillary squamous cell carcinoma and basaloid squamous cell carcinoma)
* Advanced stage but not metastatic SCC of the oral cavity (III or IVa, b); sites in the oral cavity include oral tongue, floor of mouth, hard palate, gingiva, buccal mucosa, retromolar trigone; often, head & neck tumors may involve other adjacent sites, such as the oropharynx- in these cases, the criteria is that the tumor must appear to have originated in the oral cavity per ear, nose, and throat (ENT)/radiation oncology
* Patient is deemed to be a surgical candidate by ENT
* Karnofsky performance status (KPS) 0-2
* For women of childbearing potential, a negative serum pregnancy test completed prior to any radiation therapy
* Patients with human immunodeficiency virus (HIV) infection are not automatically excluded, but must meet the following criteria: cluster of differentiation 4 (CD4) count is > 499/cu mm and their viral load is < 50 copies/ml; use of highly active antiretroviral therapy (HAART) is allowed
* Patient is free of any prior invasive malignancy (except non-melanomatous skin cancer) for a minimum of the past 3 years

Exclusion Criteria:

* Metastatic disease beyond the neck or supraclavicular area as demonstrated by positron emission tomography (PET)/CT or biopsy
* KPS 3 or worse
* Gross disease in the retrostyloid (high level II) or retropharyngeal lymph node regions by CT or PET/CT
* Patients may not have received previous therapy for their head and neck SCC, including chemotherapy, radiation therapy, or surgery beyond biopsy
* Second primary malignancy; exceptions are 1) patient had a second primary malignancy but has been treated and disease free for at least 3 years, 2) in situ carcinoma (e.g. in situ carcinoma of the cervix), 3) non-melanomatous carcinoma of the skin
* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator; this includes scleroderma
* Women who are pregnant; women of childbearing age must agree to undergo a urine pregnancy test prior to therapy and to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patient is deemed to not be a surgical candidate by ENT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional control | 2 years
  Will be assessed using both clinical and radiographic means, and recurrence will be confirmed by biopsy.

SECONDARY OUTCOMES:
Rate of pathologic complete response after preoperative hypofractionated radiation at both the primary site and lymph nodes | Up to 2 years
Rate of complete and partial response per imaging, judged per RECIST 1.1 criteria | Up to 2 years
  CT neck with IV contrast will be performed before and after radiation therapy.
Incidence of short term grade III/IV/V toxicity, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 | Up to 60 days post-surgery
  Interim analysis will be used for grade IV toxicity (death).
Incidence of long term grade III/IV/V toxicity, graded according to the NCI CTCAE, version 4.0 | Up to 2 years
Rate of flap complications (rate of flap revisions and flap complete revisions required) | Up to 2 years
Expression of molecular markers | Up to 24 hours after initial radiation treatment
  Will correlate molecular markers (especially those relating to radioresitance such as B-cell lymphoma 2 or autophagy markers to locoregional control).
Quantitative imaging characteristics in the pre-treatment PET/CT | Baseline
  Includes max/peak/total/mean standard uptake value, the metabolic tumor volume, and the total lesion glycolysis. These imaging findings will be correlated to clinical outcomes such as pathological response and locoregional control.
Changes from CT to CT (after radiation), such as changes in tumor volume or longest tumor diameter | Baseline to up to 2 years
  These imaging findings will be correlated to clinical outcomes such as pathological response and locoregional control.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Kim, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Jersey Medical School, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No